CLINICAL TRIAL: NCT04755309
Title: Electrophysiological Markers in Language and Learning Impairment: Early Intervention and Long-term Follow-up
Brief Title: Efficacy of an Early Rhythmic Intervention in Infancy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 629
Record Dates: First submitted 2021-02-05; First posted 2021-02-16 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Language Development; Language Development Disorders; Infant Development; Intervention
MeSH Terms: conditions — Language Development Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Typical development infants - experimental (Experimental): Children without familial risk for language disorders, who participate to the rhythmic intervention.
  Interventions: Behavioral: Rhythmic intervention
- Typical development infants - spontaneous development (No Intervention): No intervention is provided and typical development in children without familial risk for language disorders is evaluated.
- Typical development infants - control (Active Comparator): Children without familial risk for language disorders, who are exposed to passive auditory stimulation.
  Interventions: Behavioral: Passive auditory stimulation
- Infants at familial risk - experimental (Experimental): Children with familial risk for language disorders, who participate to the rhythmic intervention.
  Interventions: Behavioral: Rhythmic intervention
- Infants at familial risk - spontaneous development (No Intervention): No intervention is provided and typical development in children without familial risk for language disorders is evaluated.

INTERVENTIONS:
Behavioral: Rhythmic intervention — The rhythmic intervention consists in an ecological and non-invasive intervention based on enriched auditory and musical active experience. It is based on the most recent scientific evidence in the field and provides exposure to and active synchronization with complex musical rhythms. It is thought to promote the infant's ability to recognize and process the complex rhythms of spoken language. Importantly, it taps into and empowers early auditory processing skills. The intervention includes several tasks described in the literature, for example tapping and bouncing at the beat of complex musical rhythms.
  The intervention takes place in small groups of infant-caregiver pairs (N=4/5) for 1 hour/week for 6 weeks.
  Arms: Infants at familial risk - experimental; Typical development infants - experimental
Behavioral: Passive auditory stimulation — The same auditory stimulation is provided to infants, but no active tasks are proposed. Children and caregiver are entertained with motor and cognitive tasks not related to the auditory stimuli presented. The intervention takes place in small groups of infant-caregiver pairs (N=4/5) for 1 hour/week for 6 weeks.
  Arms: Typical development infants - control

SUMMARY:
The present project develops from a wide research line aiming at identifying very early electrophysiological risk markers for neurodevelopmental disorders. Long-term goals of the study include the characterization of language/learning developmental trajectories in children at high risk for language disorders and the implementation of ecological interventions based on enriched auditory experience to be employed to these children in an attempt to modify their atypical developmental trajectory before the emergence and crystallization of any behavioural symptoms and within the early period of known maximum cerebral plasticity.

Specifically, the main aim of this study is the development and implementation of an innovative and ecological early intervention based on environmental auditory enrichment (labelled "rhythmic intervention"). This intervention is tested both on a sample of typically developing infants and on a sample of infants at high familial risk for language disorders during a time span between 7 and 9 months of age. The efficacy of the intervention is tested on the electrophysiological markers tested before and after the intervention activities and on the linguistic outcomes within a longitudinal approach. The efficacy of such an intervention is compared to the spontaneous development observed in comparable groups of infants with and without familial risk for language disorders. In addition, only in a group of typically developing infants, a control intervention providing passive exposure to the same auditory stimulation is tested, in order to verify the specific contribution of the active participation of the children to the intervention.

The investigators hypothesize that the rhythmic intervention may modify the electrophysiological markers underlying auditory processing and the linguistic skills of all children, with a larger increase in infants at familial risk for language disorders who are specifically impaired in such skills.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants aged between 6 and 9 months
* Infants with and without familial risk for language disorders (Infants are assigned to the group with familial risk for language disorders if at least one first-degree relative had a certified (clinical) diagnosis of language and/or learning disorders.
* Both parents are native-Italian speakers

Exclusion Criteria:

* Gestational age < 37 weeks and/or birth-weight < 2500 grams
* APGAR scores at birth at 1' and 5' < 7
* Bayley Cognitive Score < 7
* Presence of certified diagnosis of intellectual deficiency, attention-deficit disorder, sensorial and neurological disorders or autism within first-degree relatives.

Ages: 6 Months to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 125 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Electrophysiological markers in a task tapping neural entrainment administered immediately after the end on the intervention (or at comparable age). | Age 10-11 months.
  Early neural mechanisms supporting speech and acoustic perception are recorded in response to non-speech and speech rhythmic stimuli modulated at different rates. Neural entrainment to the incoming rhythms is measured in the form of peaks emerging from the EEG spectrum at frequencies corresponding to the rhythm envelope.
Electrophysiological markers in a task tapping neural entrainment administered at age 18 months. | Age 18 months.
  Early neural mechanisms supporting speech and acoustic perception are recorded in response to non-speech and speech rhythmic stimuli modulated at different rates. Neural entrainment to the incoming rhythms is measured in the form of peaks emerging from the EEG spectrum at frequencies corresponding to the rhythm envelope.
Electrophysiological markers (obligatory peak) in a non-speech multi-feature oddball paradigm administered at age 12 months. | Age 12 months
  In the non-speech multi-feature paradigm, pairs of complex tones are presented at a rapid rate (70ms inter-stimulus interval) and stimuli differing in either frequency or duration serve as deviants. Latency of the obligatory peak (P1/P2) are computed.
Electrophysiological markers (MisMatch Response) in a non-speech multi-feature oddball paradigm administered at age 12 months. | Age 12 months
  In the non-speech multi-feature paradigm, pairs of complex tones are presented at a rapid rate (70ms inter-stimulus interval) and stimuli differing in either frequency or duration serve as deviants. Mean amplitude of the MisMatch Response is computed.
Electrophysiological markers (obligatory peak) in a non-speech multi-feature oddball paradigm administered at age 24 months. | Age 24 months
  In the non-speech multi-feature paradigm, pairs of complex tones are presented at a rapid rate (70ms inter-stimulus interval) and stimuli differing in either frequency or duration serve as deviants. Latency of the obligatory peak (P1/P2) are computed.
Electrophysiological markers (Mismatch Response) in a non-speech multi-feature oddball paradigm administered at age 24 months. | Age 24 months
  In the non-speech multi-feature paradigm, pairs of complex tones are presented at a rapid rate (70ms inter-stimulus interval) and stimuli differing in either frequency or duration serve as deviants. Mean amplitude of the MisMatch Response is computed.

SECONDARY OUTCOMES:
Expressive Language at age 12 months assessed through the Bayley Scales of Infant and Toddler Development. | Age 12 months
  Expressive language subscale of the Bayley Scales of Infant and Toddler Development. Scaled scores by age (Mean = 10, Standard Deviation = 3) are computed. Higher scores mean better performance.
Expressive Language at age 24 months assessed through the Bayley Scales of Infant and Toddler Development. | Age 24 months
  Expressive language subscale of the Bayley Scales of Infant and Toddler Development. Scaled scores by age (Mean = 10, Standard Deviation = 3) are computed. Higher scores mean better performance.
Receptive Language at age 12 months assessed through the Bayley Scales of Infant and Toddler Development. | Age 12 months
  Receptive language subscale of the Bayley Scales of Infant and Toddler Development. Scaled scores by age (Mean = 10, Standard Deviation = 3) are computed. Higher scores mean better performance.
Receptive Language at age 24 months assessed through the Bayley Scales of Infant and Toddler Development. | Age 24 months
  Receptive language subscale of the Bayley Scales of Infant and Toddler Development. Scaled scores by age (Mean = 10, Standard Deviation = 3) are computed. Higher scores mean better performance.
Expressive vocabulary at age 20 months assessed through the Language Development Survey | Age 20 months
  Number of words spontaneously produced by children, assessed through the Language Development Survey. The percentile score based on gender-specific norms is used. Higher scores mean better performance.
Expressive vocabulary at age 24 months assessed through the Language Development Survey | Age 24 months
  Number of words spontaneously produced by children, assessed through the Language Development Survey. The percentile score based on gender-specific norms is used. Higher scores mean better performance.
Mean Length Utterance assessed through the Language Development Survey | Age 24 months
  Number of words in the five longest spontaneous utterances, assessed through the Language Development Survey. The percentile score based on gender-specific norms is used. Higher scores mean better performance.
Receptive vocabulary assessed through the Picture Naming Game. | Age 20 months
  Receptive vocabulary assessed through the Picture Naming Game. The z-score based on age-specific norms is used (Mean = 0, Standard Deviation = 1). Higher scores mean better performance.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Eugenio Medea, Bosisio Parini, LC, Italy

IPD SHARING:
Plan to Share IPD: No